CLINICAL TRIAL: NCT00003646
Title: Phase II Study of Allovectin-7 as an Immunotherapeutic Agent in Patients With Stages III and IV Melanoma
Brief Title: Gene Therapy in Treating Patients With Stage III or Stage IV Melanoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Vical (Industry)
Responsible Party: Dmitri D. Kharkevitch, MD, PhD, Vical Incorporated
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000066735; VCL-1005-205 (Other: Vical); NCT00416806 (obsolete NCT alias)
Record Dates: First submitted 1999-11-01; First posted 2004-05-03 (Estimated); Last update posted 2011-07-07 (Estimated); Status verified 2011-07

CONDITIONS: Stage IV Melanoma; Stage III Melanoma; Recurrent Melanoma
Keywords: adult solid tumor; body system/site cancer; cancer; melanoma; recurrent melanoma; skin tumor; solid tumor; stage III melanoma; stage IV melanoma; stage, melanoma
MeSH Terms: conditions — Melanoma; Neoplasms; Skin Neoplasms | interventions — Allovectin-7

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Drug: allovectin-7

SUMMARY:
RATIONALE: Injecting allovectin-7 into a person's melanoma cells may make the body build an immune response that will kill tumor cells.

PURPOSE: Phase II trial to study the effectiveness of gene therapy in treating patients who have stage III or stage IV melanoma that has not responded to previous treatment.

DETAILED DESCRIPTION:
OBJECTIVES: I. Demonstrate an objective clinical response (partial or complete) with a median duration of at least 4 months in 15% of patients with stage III or IV melanoma treated with Allovectin-7. Allovectin-7 is a direct gene transfer immunotherapeutic agent.

II. Determine the benefits, risks, and side effects of Allovectin-7 in this patient population.

PROTOCOL OUTLINE: This is a multicenter study. Patients receive an intratumoral injection of Allovectin-7 once weekly for 6 weeks. At week 9, a complete disease status assessment is performed. Patients with stable or responding disease may receive additional courses of 6 injections.

PROJECTED ACCRUAL:

A total of 70 patients will be accrued for this study.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Histologically confirmed melanoma; Stage III with locoregional disease, in transit metastasis, or nodal disease OR Stage IV metastatic disease in skin, subcutaneous tissue, lymph node(s), and/or lung
* At least 1 metastasis for which surgery is not deemed to be a curative option
* Relapsed from or has not responded to frontline chemotherapy or biotherapy
* At least 1 measurable tumor at least 1 cm by 1 cm, but less than 5 cm by 5 cm
* No history of brain metastases or visceral metastases other than lung metastases

--Prior/Concurrent Therapy--

* Biologic therapy: See Disease Characteristics; At least 4 weeks since prior biologic therapy
* Chemotherapy: See Disease Characteristics; At least 4 weeks since prior chemotherapy
* Endocrine therapy: No concurrent immunosuppressive drugs
* Radiotherapy: At least 4 weeks since prior radiotherapy
* Surgery: At least 2 weeks since prior major surgery
* Other: No other concurrent anticancer drug therapy, or any other experimental therapy

--Patient Characteristics--

* Age: 18 and over
* Performance status: Karnofsky 80-100%
* Life expectancy: At least 6 months
* Hematopoietic: WBC at least 3,000/mm3; Platelet count at least 100,000/mm3; Hemoglobin at least 9 g/dL
* Hepatic: Bilirubin no greater than 2.0 mg/dL; SGOT/SGPT less than 3 times upper limit of normal; PT/PTT normal LDH and albumin normal
* Renal: Creatinine no greater than 2.0 mg/dL
* Cardiovascular: No uncontrolled hypertension; No New York Heart Association class III or IV disease
* Other: HIV negative; Negative pregnancy test; Fertile patients must use effective contraception; No active autoimmune disease; No active infection requiring parenteral antibiotics; No uncontrolled diabetes mellitus; No other prior malignancy in the past 5 years except skin cancer or stage 0-II cervical cancer; No significant psychiatric disorders

Min Age: 18 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 78 (Actual)
Dates: Start 1998-08; Primary Completion 2002-03 (Actual); Study Completion 2002-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer Fernandez, Study Chair — Vical
Locations (3):
- United States (3):
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Roswell Park Cancer Institute, Buffalo, New York
  - Physician Reliance Network, Inc., Dallas, Texas